CLINICAL TRIAL: NCT03580590
Title: Efficacy of Oral Diltiazem Versus Combination of Oral Diltiazem With Intravenous Tranexamic Acid on the Intraoperative Bleeding in Functional Endoscopic Sinus Surgery
Brief Title: Efficacy of Oral Diltiazem on the Intraoperative Bleeding in Functional Endoscopic Sinus Surgery
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Moutaz Ragab Ismail Ibrahim, M.D, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: Oral diltiazem in FESS
Record Dates: First submitted 2018-06-12; First posted 2018-07-09 (Actual); Last update posted 2018-07-09 (Actual); Status verified 2018-06

CONDITIONS: Hypotension on Induction
MeSH Terms: interventions — Diltiazem; Tranexamic Acid; capron

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- 1st group (Experimental): 20 patients will receive 90 mg oral Diltiazem 3 hours pre-operative
  Interventions: Drug: oral Diltiazem
- 2nd group (Experimental): 20 patients will receive 90 mg oral Diltiazem 3 hours pre-operative+ 10 mg/kg IV Tranexamic Acid slow infusion with saline half an hour before the induction of anesthesia
  Interventions: Drug: oral Diltiazem; Drug: IV Tranexamic Acid
- 3rd group (Placebo Comparator): 20 patients will receive oral placebo tablet 3 hours pre-operative
  Interventions: Drug: Placebo Oral Tablet

INTERVENTIONS:
Drug: oral Diltiazem — Diltiazem, a calcium channel blocker reduced arteriolar tone and fall in blood pressure
  Other Names: diltiazem
  Arms: 1st group; 2nd group
Drug: IV Tranexamic Acid — Tranexamic acid inhibits fibrinolysis, which reduces blood loss
  Other Names: capron
  Arms: 2nd group
Drug: Placebo Oral Tablet — Placebo Oral Tablet
  Arms: 3rd group

SUMMARY:
* The primary endpoint is the effect of the addition of oral Diltiazem and Tranexamic Acid to general anesthesia aided reduction in blood loss during functional endoscopic sinus surgery (FESS).
* The secondary endpoint is surgeon's assessment of the surgical field and hemodynamics.

DETAILED DESCRIPTION:
Functional endoscopic sinus surgery (FESS) is a minimally invasive technique used to restore sinus ventilation and function in patients with recurrent acute or chronic infective sinusitis in whom medical therapy has failed.

Continued bleeding into the surgical field during FESS not only impairs endoscopic vision but can lead to complications.

Controlled hypotension is a technique used to limit intraoperative blood loss to provide the best possible field for surgery. The physiological principle which underlies hypotensive anesthesia is a natural survival mechanism. When profuse bleeding occurs, the blood pressure drops. This drop leads to a reduction or cessation of the bleeding, blood pressure stabilization, and recovery. Accordingly, reducing the patient's blood pressure during surgery can potentially reduce overall bleeding. Since bleeding in the surgical field is also reduced, the surgical field operating conditions are improved In hypotensive anesthesia, the patient's baseline mean arterial pressure (MAP) is reduced by 30 %. Consequently, the systolic blood pressure values are about 80-90mmHg and the MAP is reduced to 50- 65mmHg.

Hypotensive anesthesia is considered to be a suitable anesthetic technique for those patients who will be undergoing spinal surgery, hip or knee arthroplasty, craniosynostosis, hepatic resections, and major maxillofacial operations. Benefits for controlled hypotension for FESS include the reduction in blood loss with improved quality of the surgical field.

Various agent's anesthetic agents, analgesics, and hypotensive drugs, that have been used for achieving hypotensive anesthesia:

1. Volatile Anesthetic Agents. Most anesthetic agents have a hypotensive effect such as isoflurane, sevoflurane, and desflurane, high concentrations are required to achieve a significant reduction in intraoperative bleeding, and these concentrations may lead to hepatic or renal injury.
2. Propofol. has a potent hypotensive capability, but normal blood pressure will be rapidly restored when the propofol infusion is discontinued. Although a short-term propofol infusion is safe, a long-term Propofol infusion can cause propofol infusion syndrome in children.
3. Alfentanil, Sufentanil, and Remifentanil. potent synthetic and short-acting opioid drugs, Since the recovery times from this type of anesthesia are also short, they are widely used for hypotensive anesthesia.

d.Nitrates. SNP and NTG are two very potent hypotensive agents that are commonly used for inducing hypotensive anesthesia. Reflex tachycardia is an unwanted effect which often occurs with nitrates administration and can be prevented by a small dose of the beta-adrenoceptor antagonist, such as esmolol or propranolol premedication.

e-beta-Adrenoceptor Antagonists. They effectively used for inducing hypotensive anesthesia when administered either as a single hypotensive agent or in combination with SNP. Nonselective beta-antagonists, such as labetalol, may cause bronchoconstriction and should be avoided in asthmatic patients. The hypotensive action of beta-adrenoceptor antagonists is achieved by reducing cardiac output. So, not suitable for the patient with underlying heart failure.

f-Calcium Channel Antagonists. such as nifedipine or nicardipine, are commonly used as hypotensive drugs.

Diltiazem, a calcium channel blocker, blocks the influx of calcium into smooth muscle cells and cardiac muscle cells. This causes relaxation of the muscle, thereby causing reduced arteriolar tone and fall in blood pressure.

Tranexamic acid is a synthetic amino acid that inhibits fibrinolysis, which reduces blood loss and the need for blood transfusion in total knee arthroplasty, spine surgery, and cardiac surgery. It has seen wide application in a variety of surgical procedures since then.

ELIGIBILITY:
Inclusion Criteria:

include patients who undergoing elective FESS under general anesthesia and meet these criteria:

- Age from 18 - 60 years old. - ASA grade I - II.

Exclusion Criteria:

* - Patient refusal.
* Any contraindication of calcium channel blocker:

  1. AV conduction defects (2nd and 3rd degree AV block).
  2. Sick sinus syndrome.
  3. Wolf-Parkinson-White Syndrome.
  4. History of congestive heart failure.
  5. Patients on long-term ß-blocker therapy.
* Patients with allergy to medication included in the study.
* Any contraindication of Tranexamic Acid:

  1. bleeding disorders.
  2. pregnant or breastfeeding mothers.
  3. patient under the influence of anticoagulants.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2018-09-01 (Estimated); Primary Completion 2019-11-01 (Estimated); Study Completion 2020-01-01 (Estimated)

PRIMARY OUTCOMES:
Estimated Blood Loss | end of operation assessment
  Estimated blood loss in milliliters per hour is calculated by subtracting the volume of total irrigation used during the case from the total amount of fluid in the suction canister at the end of surgery dividing by surgical time in hours.

SECONDARY OUTCOMES:
The Boezaart and van der Merwe intraoperative surgical field scale | Every 15 minutes for the duration of surgery
  Boezaart Bleeding Scale (BBS) (0 - no bleeding (cadaveric conditions), 1 - Slight bleeding, no suctioning required, 2 - Slight bleeding, occasional suctioning required, 3 - Slight bleeding, frequent suctioning required; bleeding threatens surgical field a few seconds after suction is removed, 4 - Moderate bleeding, frequent suctioning required, and bleeding threatens surgical field directly after suction is removed, 5 - Severe bleeding, constant suctioning required; bleeding appears faster than can be removed by suction; surgical field severely threatened and surgery usually not possible).
Incidence of hypotension | Hemodynamic parameters as systolic, diastolic and mean arterial blood pressures were recorded before drug intake, before induction, after induction, intraoperative every 5 minutes till the end of surgery, every 15 minutes post operative
  systolic blood pressure values are 80-90mmHg Mean arterial pressure is reduced to 50-65mmHg
total consumption of propofol | end of operation assessment
  The investigators will measure the consumption of propofol intraoperatively
Heart Rate | Heart Rate recorded before drug intake, before induction, after induction, intraoperative every 5 minutes till the end of surgery, every 15 minutes postoperative
  heart beats for minutes
End Tidal CO2 | End Tidal CO2 before induction, after induction, intraoperative every 5 minutes till the end of surgery
  The concentration of carbon dioxide (CO2) in the respiratory gases

CONTACTS AND LOCATIONS:
Overall Officials: Hamdy Abbas Youssef, PhD, Study Director — Assiut Univerity

REFERENCES:
- [Background] Aravindan A, Subramanium R, Chhabra A, Datta PK, Rewari V, Sharma SC, Kumar R. Magnesium sulfate or diltiazem as adjuvants to total intravenous anesthesia to reduce blood loss in functional endoscopic sinus surgery. J Clin Anesth. 2016 Nov;34:179-85. doi: 10.1016/j.jclinane.2016.03.068. Epub 2016 May 10. PMID 27687369